CLINICAL TRIAL: NCT07191886
Title: Measuring Patient Reported Needs in Outpatient Liver Disease Management
Status: Recruiting | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Archita P. Desai, Assistant Professor of Medicine, Indiana University
Other Study IDs: PRN Study
Record Dates: First submitted 2025-09-17; First posted 2025-09-25 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Chronic Liver Disease; Cirrhosis, Liver
Keywords: health-related social needs; social determinants of health; patient-reported outcomes; quality of life
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with Chronic Liver Disease: Adults (≥18 years) with chronic liver disease receiving outpatient care in hepatology clinics at Indiana University Health University Hospital. Participants will complete surveys assessing health-related social needs, health literacy, quality of life, social support, patient activation, and technology use. Relevant demographic, medical history, and clinical data will also be abstracted from the electronic medical record.
- Outpatient Liver Care Providers: Healthcare providers (physicians, nurse practitioners, physician assistants, or other clinical staff) who deliver care to enrolled patients during study visits. Providers will complete a survey regarding their experiences with health-related social needs screening and perspectives on how this information might be integrated into routine practice.

SUMMARY:
This prospective study aims to assess health-related social needs (HRSNs) among patients with chronic liver disease (CLD) receiving outpatient care at Indiana University Health. Patients with CLD often face socioeconomic challenges that adversely affect health outcomes, but no validated screening tool exists for this population. The primary objective is to measure the prevalence and types of HRSNs in CLD patients. Secondary objectives are to evaluate patient preferences regarding provider involvement in addressing social needs, explore reasons for declining assistance, and assess provider perspectives on incorporating HRSN data into clinical care.

A total of 200 adult patients with CLD and their visit providers will be enrolled. Participants will complete surveys on demographics, HRSNs, health literacy, quality of life, social support, and patient activation, with medical data supplemented from chart review. Providers will complete surveys about their experiences using HRSN data in routine practice. Results will describe unmet social needs in this population, patient and provider attitudes toward screening, and inform strategies for integrating HRSN assessments into liver disease management and routine healthcare delivery.

DETAILED DESCRIPTION:
Patients with chronic liver disease (CLD) are a medically and socially vulnerable population who often face significant health-related social needs (HRSNs), such as financial strain, housing instability, limited access to transportation, and lack of social support. These unmet needs contribute to poorer health outcomes and higher healthcare utilization, yet there is currently no validated screening tool specifically designed for patients with CLD. In addition, little is known about whether patients want their healthcare providers to address these needs, or how providers might use such information in routine practice.

This study is designed to measure the prevalence of HRSNs in patients with CLD receiving care in outpatient liver clinics, and to explore patient and provider perspectives on the role of HRSN screening in clinical care. Patients will complete surveys assessing HRSNs, health literacy, quality of life, social support, and patient activation, with additional demographic and clinical information obtained from chart review. Providers will complete surveys regarding their experience and potential use of HRSN data.

By combining patient- and provider-reported data, this study will generate new insights into the burden of unmet social needs in CLD, patient preferences for assistance from their care team, and provider attitudes toward incorporating HRSN data into clinical management. Findings are expected to inform the development and implementation of standardized HRSN screening approaches in liver disease care, with the broader goal of improving patient-centered outcomes and aligning with evolving healthcare quality standards.

ELIGIBILITY:
Inclusion Criteria:

* Patient Inclusion criteria

  * Age 18 or greater
  * English speaking
  * Ability to give consent (West Haven stage 0-1 if history of hepatic encephalopathy)

Provider Inclusion Criteria • Participated in patient care during inclusion visit

Exclusion Criteria:

* Patient Exclusion criteria

  * History of liver transplant
  * Individuals not willing to participate in the survey
  * Patients with severe cognitive impairment

Provider Exclusion Criteria

• Unable to complete survey within 7 days of the inclusion visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with chronic liver disease receiving outpatient care in hepatology clinics at Indiana University Health University Hospital and providers delivering care during the study visits.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence and Types of Health-Related Social Needs (HRSNs) | Day 1
  Proportion and categories of health-related social needs reported by patients with chronic liver disease using a structured HRSN survey.

SECONDARY OUTCOMES:
Patient Preferences for Provider Involvement in Addressing HRSNs | Day 1
  Proportion of patients who indicate they would like their liver care team to assist with addressing identified social needs, as measured by survey responses.
Reasons Patients Decline Provider Assistance with HRSNs | Day 1
  Reported reasons why patients prefer not to seek provider assistance with social needs, captured through structured survey items.
Provider Perspectives on HRSN Screening | Within 7 days of patient visit
  Provider-reported attitudes and experiences with HRSN screening, including perceived usefulness and likelihood of incorporating results into clinical care, as measured by provider survey.
Association Between HRSNs and Clinical Characteristics | Day 1, with retrospective chart review (12 months prior healthcare utilization and labs)
  Relationship between reported HRSNs and clinical factors such as comorbidities, liver disease etiology, hospitalizations, ED visits, and MELD-Na score, using statistical correlation analyses.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No